CLINICAL TRIAL: NCT01350843
Title: An Investigation Into the Effects of Orange Juice on Plasma Lipids - an Extension to J/06/2010
Brief Title: The Effects of Orange Juice on Plasma Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Florida Department of Citrus (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RIS 100058b
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Insulin Resistance; Obesity; Dyslipidemia
Keywords: Men; Orange Juice; Cholesterol; Obesity
MeSH Terms: conditions — Insulin Resistance; Obesity; Dyslipidemias; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orange Juice (Experimental): Juice high in flavonoids
  Interventions: Dietary Supplement: Orange Juice
- Orange Drink (Placebo Comparator): Sugars matched, low flavonoids orange drink
  Interventions: Dietary Supplement: Orange Juice

INTERVENTIONS:
Dietary Supplement: Orange Juice — 250ml of orange juice or a sugars matched orange drink daily

SUMMARY:
The aim of this study is primarily to investigate the ability of antioxidants found in orange juice (OJ) to improve the serum lipid profile. Overweight or mildly obese men, who are otherwise healthy, but with elevated serum total cholesterol concentration will be recruited. The time commitment for subjects is ~14wks. Subjects will attend the laboratory on 5 occasions after fasting from midnight. The 1st is a medical screening. Laboratory visits 2 & 5 will take ~90min and will be separated by 3 months, during which time subjects will consume 250ml of an orange drink (either OJ or an orange flavoured control drink) once a day. During visits 2 & 5, subjects will have a scan to assess their %body fat using a low-dose x-ray machine, a 20ml blood sample taken and a small sample of fat tissue (about the size of a haricot bean)taken from underneath the skin of the belly. Subjects will record their food intake for 3-days in weeks 3, 7 and 11 of consuming the drink, and come to the lab for visits 3&4 during weeks 4&8. Laboratory visits 3&4 repeat measurements taken in the 1st (screening) visit.

DETAILED DESCRIPTION:
Background:

Overweight and mild obesity are associated with insulin resistance and mild elevations in lipid risk factors which are not usually sufficiently abnormal to merit treatment. Such people are encouraged to lose weight to reduce their risk of progressing to type 2 diabetes and coronary heart disease, but there is clearly a potential role for dietary modifications to maximize any potential benefit of this weight loss. Flavonoids are known to have vascular effects which might enhance substrate delivery to metabolically active tissues, and thus improve insulin sensitivity. Moreover, there is much interest in the potentially beneficial effect of flavonoids on serum lipid profile.

There are many different dietary sources of flavonoids, with fruits such as apples, berries and citrus being rich sources. However, some researchers have expressed concern that a high dietary intake of 100% juice may contribute to the development of insulin resistance, obesity and the Metabolic Syndrome (Bazzano, Li et al. 2008), although this is not universally accepted (Fujioka, Greenway et al. 2006; O'Neil and Nicklas 2008). To date, there have been no studies investigating the effects of citrus fruits on indices of cardio-metabolic health in people who are presently healthy but are at risk of developing some features of the Metabolic Syndrome.

Aims:

To investigate the effects of orange juice (OJ) intake on appetite hormones, blood pressure and plasma lipids. In addition we aim to investigate any gene expression changes associated with OJ consumption, in particular in adipose tissue.

Experimental protocol and methods:

Overweight or obese men (BMI 27-35), who are otherwise healthy, will be recruited onto the study. They will attend the 'David Greenfield Human Physiology' laboratories on 5 convenient mornings, following an overnight fast. The 1st visit is a medical screening and will involve signing a consent form, completing medical screening, food frequency and activity questionnaires, having height, weight, and hip/waist circumference measurements taken and a sample of blood taken for CBC, urea, electrolytes, LFT, TFT, glucose and insulin analysis. Subjects will then be asked to complete a 3-day diet diary for macronutrient assessment. The 2nd visit will involve having a DEXA body composition scan, an adipose tissue biopsy and a blood sample taken for white blood cell harvest, serum lipids, glucose, insulin, cytokines, appetite hormones and catecholamine analysis. Starting on the following morning, subjects will then consume an orange drink (either OJ or a carbohydrate matched orange flavoured drink) once a day for 12 wks. A 3-day diet diary for macronutrient assessment will be recorded during wks 3,7and 11 of taking the drink, and measurements made at screening will be repeated on visits 3 and 4 which will take place in weeks 4 and 8. The final laboratory (5th) visit will be identical to visit 2.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-35
* waist circumference >96cm.
* Serum Total Cholesterol >5mmol/l

Exclusion Criteria:

* Any clinically significant metabolic or endocrine abnormalities
* screening blood results (other than lipids) outside of the normal range
* fasting total cholesterol >7.0mmol/l
* taking routine medication
* herbal supplement use
* food allergies or sensitivities related to the investigational product Regular citrus consumers (whole fruit or juice) daily consumption of sucrose or high fructose corn syrup containing soft-drinks

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Total Serum Cholesterol concentration | after 3 months' intervention
  Fasting Serum total cholesterol concentration (mmol/l)

SECONDARY OUTCOMES:
High Density Cholesterol (HDL) | after 3 months' intervention
  Fasting Serum HDL concentration
Low density cholesterol | after 3 months' intervention
  Fasting Serum LDL concentration
Gene expression in adipose tissue | after 3 months' intervention
  Expression of genes related to lipid metabolism in adipose tissue
leptin | after 3 month intervention
  fasting Serum Leptin concentration
IL-1 | afetr 3 month intervention
  Serum IL-1 concentration
Blood Pressure | after 3months intervention
  Resting blood pressure, measured semi-supine
Ghrelin | After 3 months intervention
  Fasting Plasma Ghrelin concentration
GLP-1 | After 3 months intervention
  Fasting Plasma GLP-1 concentration
insulin | After 3 months intervention
  Fasting serum Insulin concentration
IL-6 | After 3 months intervention
  Serum IL-6 concentration
TNF alpha | After 3 months intervention
  Serum TNF-Alpha concentration

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Macdonald, PhD, Principal Investigator — Nottingham University
Locations (1):
- David Greenfield Human Physiology Unit, University of Nottingham, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bazzano LA, Li TY, Joshipura KJ, Hu FB. Intake of fruit, vegetables, and fruit juices and risk of diabetes in women. Diabetes Care. 2008 Jul;31(7):1311-7. doi: 10.2337/dc08-0080. Epub 2008 Apr 4. PMID 18390796
- [Background] Fujioka K, Greenway F, Sheard J, Ying Y. The effects of grapefruit on weight and insulin resistance: relationship to the metabolic syndrome. J Med Food. 2006 Spring;9(1):49-54. doi: 10.1089/jmf.2006.9.49. PMID 16579728
- [Background] O'Neil CE, Nicklas TA. A review of the relationship between 100% fruit juice consumption and weight in children and adolescents. American Journal of Lifestyle Medicine 2(4): 315-354, 2008.
- [Result] Simpson EJ, Mendis B, Macdonald IA. Orange juice consumption and its effect on blood lipid profile and indices of the metabolic syndrome; a randomised, controlled trial in an at-risk population. Food Funct. 2016 Apr;7(4):1884-91. doi: 10.1039/c6fo00039h. PMID 26965492